CLINICAL TRIAL: NCT07224802
Title: An Exosome-based Liquid Biopsy Signature for Preoperative Identification of Occult Liver Metastasis in Patients With Pancreatic Ductal Adenocarcinoma
Brief Title: Forecasting Occult liveR Metastasis Using an Exosomal Signature for Intelligent Guided Hepatic Targeting
Acronym: FORESIGHT
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19288/FORESIGHT
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: pancreatic ductal adenocarcinoma; exosomal miRNA; early liver metastasis; liquid biopsy; exosome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Training Cohort - PDAC with Occult Liver Metastasis: Patients with PDAC who were found to have occult liver metastases at the time of or shortly after curative-intent pancreatectomy (within 6 months post-surgery), in the first cohort (training set).
  Interventions: Diagnostic Test: EXELiM assay (qRT-PCR validation)
- Training Cohort - PDAC without Occult Liver Metastasis: Patients with PDAC who did not develop liver metastasis for at least 6 months after curative-intent surgery in the first cohort (training set).
  Interventions: Diagnostic Test: EXELiM assay (qRT-PCR validation)
- Validation Cohort - PDAC with Occult Liver Metastasis: Patients with PDAC who were found to have occult liver metastases (early postoperative hepatic recurrence within 6 months) in the second cohort (validation set).
  Interventions: Diagnostic Test: EXELiM assay (qRT-PCR validation)
- Validation Cohort - PDAC without Occult Liver Metastasis: Patients with PDAC who did not develop liver metastasis for at least 6 months after curative-intent surgery in the second cohort (validation set).
  Interventions: Diagnostic Test: EXELiM assay (qRT-PCR validation)
- Discovery Cohort - PDAC with Occult Liver Metastasis: Patients with PDAC who were found to have occult liver metastases at the time of or shortly after curative-intent pancreatectomy (within 6 months post-surgery), in the discovery cohort.
  Interventions: Diagnostic Test: EXELiM small RNA sequencing
- Discovery Cohort - PDAC without Occult Liver Metastasis: Patients with PDAC who did not develop liver metastasis for at least 6 months after curative-intent surgery in the discovery cohort.
  Interventions: Diagnostic Test: EXELiM small RNA sequencing

INTERVENTIONS:
Diagnostic Test: EXELiM assay (qRT-PCR validation) — Quantitative reverse-transcription PCR (qRT-PCR)-based validation assay performed on preoperative plasma samples from PDAC patients in the training and validation cohorts.
  Candidate microRNAs identified by small RNA sequencing were tested using the EXELiM assay to validate their predictive accuracy for occult liver metastasis detection prior to surgery.
  Groups: Training Cohort - PDAC with Occult Liver Metastasis; Training Cohort - PDAC without Occult Liver Metastasis; Validation Cohort - PDAC with Occult Liver Metastasis; Validation Cohort - PDAC without Occult Liver Metastasis
Diagnostic Test: EXELiM small RNA sequencing — High-throughput small RNA sequencing performed on preoperative plasma samples from PDAC patients in the discovery cohort to identify exosome-derived microRNAs associated with occult liver metastasis or early postoperative hepatic recurrence.
  Groups: Discovery Cohort - PDAC with Occult Liver Metastasis; Discovery Cohort - PDAC without Occult Liver Metastasis

SUMMARY:
Early liver metastasis (Early-LiM) is the most significant prognostic factor in pancreatic ductal adenocarcinoma (PDAC) and is thought to originate from occult micrometastases present at the time of surgery. Reliable preoperative detection of such lesions remains an unmet clinical need.

The EXELiM study aims to develop and validate a circulating exosomal microRNA (exo-miRNA)-based liquid biopsy assay to accurately identify PDAC patients at high risk of occult liver metastasis before surgery. By integrating machine learning with multi-institutional plasma exosome profiling, this study seeks to enable biology-driven patient stratification and guide treatment sequencing toward precision oncology.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is one of the deadliest human malignancies, with a 5-year overall survival rate below 10%. Even after curative-intent pancreatectomy, over 70% of patients experience disease recurrence, with early liver metastasis (within six months postoperatively) representing the most aggressive and fatal pattern.

Emerging evidence indicates that pancreatic tumors release exosomes that modulate the liver microenvironment, establishing a premetastatic niche that facilitates early colonization. We hypothesize that circulating exosomal microRNAs reflect these biological processes and can serve as non-invasive biomarkers for detecting occult liver metastasis.

In this multi-center observational study, preoperative plasma-derived exosomes from PDAC patients are analyzed using next-generation small RNA sequencing and validated by RT-qPCR. A machine learning model is employed to integrate exo-miRNA expression profiles and clinical variables, yielding a predictive score for early liver metastasis risk.

The study evaluates the diagnostic accuracy, prognostic utility, and clinical benefit of the exo-miRNA panel compared to conventional biomarkers such as CA19-9.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic ductal adenocarcinoma (PDAC)
* Undergoing curative-intent pancreatectomy
* Availability of preoperative plasma samples
* Complete clinical and follow-up data
* Written informed consent obtained

Exclusion Criteria:

* Synchronous or secondary malignancies
* Non-adenocarcinoma histology
* Lack of informed consent
* Incomplete plasma sample data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed pancreatic ductal adenocarcinoma (PDAC) who have undergone curative-intent pancreatectomy with available preoperative plasma samples.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Specificity | Through study completion, an average of 3 year
  True Negative Rate: probability of a negative test result conditioned on absence of early liver metastasis

SECONDARY OUTCOMES:
Sensitivity | Through study completion, an average of 3 year
  True Positive Rate: probability of a positive test result conditioned on the presence of early liver metastasis
Area Under the Receiver Operating Characteristic Curve (AUC) | Through study completion, an average of 3 year
  Description: AUC representing the overall discriminative ability of the circRNA-based model.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data.

REFERENCES:
- [Background] Costa-Silva B, Aiello NM, Ocean AJ, Singh S, Zhang H, Thakur BK, Becker A, Hoshino A, Mark MT, Molina H, Xiang J, Zhang T, Theilen TM, Garcia-Santos G, Williams C, Ararso Y, Huang Y, Rodrigues G, Shen TL, Labori KJ, Lothe IM, Kure EH, Hernandez J, Doussot A, Ebbesen SH, Grandgenett PM, Hollingsworth MA, Jain M, Mallya K, Batra SK, Jarnagin WR, Schwartz RE, Matei I, Peinado H, Stanger BZ, Bromberg J, Lyden D. Pancreatic cancer exosomes initiate pre-metastatic niche formation in the liver. Nat Cell Biol. 2015 Jun;17(6):816-26. doi: 10.1038/ncb3169. Epub 2015 May 18. PMID 25985394
- [Background] Hoshino A, Costa-Silva B, Shen TL, Rodrigues G, Hashimoto A, Tesic Mark M, Molina H, Kohsaka S, Di Giannatale A, Ceder S, Singh S, Williams C, Soplop N, Uryu K, Pharmer L, King T, Bojmar L, Davies AE, Ararso Y, Zhang T, Zhang H, Hernandez J, Weiss JM, Dumont-Cole VD, Kramer K, Wexler LH, Narendran A, Schwartz GK, Healey JH, Sandstrom P, Labori KJ, Kure EH, Grandgenett PM, Hollingsworth MA, de Sousa M, Kaur S, Jain M, Mallya K, Batra SK, Jarnagin WR, Brady MS, Fodstad O, Muller V, Pantel K, Minn AJ, Bissell MJ, Garcia BA, Kang Y, Rajasekhar VK, Ghajar CM, Matei I, Peinado H, Bromberg J, Lyden D. Tumour exosome integrins determine organotropic metastasis. Nature. 2015 Nov 19;527(7578):329-35. doi: 10.1038/nature15756. Epub 2015 Oct 28. PMID 26524530
- [Background] Bojmar L, Zambirinis CP, Hernandez JM, Chakraborty J, Shaashua L, Kim J, Johnson KE, Hanna S, Askan G, Burman J, Ravichandran H, Zheng J, Jolissaint JS, Srouji R, Song Y, Choubey A, Kim HS, Cioffi M, van Beek E, Sigel C, Jessurun J, Velasco Riestra P, Blomstrand H, Jonsson C, Jonsson A, Lauritzen P, Buehring W, Ararso Y, Hernandez D, Vinagolu-Baur JP, Friedman M, Glidden C, Firmenich L, Lieberman G, Mejia DL, Nasar N, Mutvei AP, Paul DM, Bram Y, Costa-Silva B, Basturk O, Boudreau N, Zhang H, Matei IR, Hoshino A, Kelsen D, Sagi I, Scherz A, Scherz-Shouval R, Yarden Y, Oren M, Egeblad M, Lewis JS, Keshari K, Grandgenett PM, Hollingsworth MA, Rajasekhar VK, Healey JH, Bjornsson B, Simeone DM, Tuveson DA, Iacobuzio-Donahue CA, Bromberg J, Vincent CT, O'Reilly EM, DeMatteo RP, Balachandran VP, D'Angelica MI, Kingham TP, Allen PJ, Simpson AL, Elemento O, Sandstrom P, Schwartz RE, Jarnagin WR, Lyden D. Multi-parametric atlas of the pre-metastatic liver for prediction of metastatic outcome in early-stage pancreatic cancer. Nat Med. 2024 Aug;30(8):2170-2180. doi: 10.1038/s41591-024-03075-7. Epub 2024 Jun 28. PMID 38942992
- [Background] Tang D, Wang D, Yuan Z, Xue X, Zhang Y, An Y, Chen J, Tu M, Lu Z, Wei J, Jiang K, Miao Y. Persistent activation of pancreatic stellate cells creates a microenvironment favorable for the malignant behavior of pancreatic ductal adenocarcinoma. Int J Cancer. 2013 Mar 1;132(5):993-1003. doi: 10.1002/ijc.27715. Epub 2012 Oct 5. PMID 22777597
- [Background] Grunwald B, Harant V, Schaten S, Fruhschutz M, Spallek R, Hochst B, Stutzer K, Berchtold S, Erkan M, Prokopchuk O, Martignoni M, Esposito I, Heikenwalder M, Gupta A, Siveke J, Saftig P, Knolle P, Wohlleber D, Kruger A. Pancreatic Premalignant Lesions Secrete Tissue Inhibitor of Metalloproteinases-1, Which Activates Hepatic Stellate Cells Via CD63 Signaling to Create a Premetastatic Niche in the Liver. Gastroenterology. 2016 Nov;151(5):1011-1024.e7. doi: 10.1053/j.gastro.2016.07.043. Epub 2016 Aug 6. PMID 27506299
- [Background] Houg DS, Bijlsma MF. The hepatic pre-metastatic niche in pancreatic ductal adenocarcinoma. Mol Cancer. 2018 Jun 14;17(1):95. doi: 10.1186/s12943-018-0842-9. PMID 29903049
- [Background] Lee JW, Stone ML, Porrett PM, Thomas SK, Komar CA, Li JH, Delman D, Graham K, Gladney WL, Hua X, Black TA, Chien AL, Majmundar KS, Thompson JC, Yee SS, O'Hara MH, Aggarwal C, Xin D, Shaked A, Gao M, Liu D, Borad MJ, Ramanathan RK, Carpenter EL, Ji A, de Beer MC, de Beer FC, Webb NR, Beatty GL. Hepatocytes direct the formation of a pro-metastatic niche in the liver. Nature. 2019 Mar;567(7747):249-252. doi: 10.1038/s41586-019-1004-y. Epub 2019 Mar 6. PMID 30842658
- [Background] Chikhladze S, Lederer AK, Kousoulas L, Reinmuth M, Sick O, Fichtner-Feigl S, Wittel UA. Adjuvant chemotherapy after surgery for pancreatic ductal adenocarcinoma: retrospective real-life data. World J Surg Oncol. 2019 Nov 9;17(1):185. doi: 10.1186/s12957-019-1732-3. PMID 31706323
- [Background] Merkow RP, Bilimoria KY, Tomlinson JS, Paruch JL, Fleming JB, Talamonti MS, Ko CY, Bentrem DJ. Postoperative complications reduce adjuvant chemotherapy use in resectable pancreatic cancer. Ann Surg. 2014 Aug;260(2):372-7. doi: 10.1097/SLA.0000000000000378. PMID 24374509
- [Background] Powell-Brett S, Pande R, Roberts KJ. Achieving 'Marginal Gains' to Optimise Outcomes in Resectable Pancreatic Cancer. Cancers (Basel). 2021 Apr 1;13(7):1669. doi: 10.3390/cancers13071669. PMID 33916294
- [Background] Zambirinis CP, Midya A, Chakraborty J, Chou JF, Zheng J, McIntyre CA, Koszalka MA, Wang T, Do RK, Balachandran VP, Drebin JA, Kingham TP, D'Angelica MI, Allen PJ, Gonen M, Simpson AL, Jarnagin WR. Recurrence After Resection of Pancreatic Cancer: Can Radiomics Predict Patients at Greatest Risk of Liver Metastasis? Ann Surg Oncol. 2022 Aug;29(8):4962-4974. doi: 10.1245/s10434-022-11579-0. Epub 2022 Apr 3. PMID 35366706
- [Background] Seelen LWF, Floortje van Oosten A, Brada LJH, Groot VP, Daamen LA, Walma MS, van der Lek BF, Liem MSL, Patijn GA, Stommel MWJ, van Dam RM, Koerkamp BG, Busch OR, de Hingh IHJT, van Eijck CHJ, Besselink MG, Burkhart RA, Borel Rinkes IHM, Wolfgang CL, Molenaar IQ, He J, van Santvoort HC. Early Recurrence After Resection of Locally Advanced Pancreatic Cancer Following Induction Therapy: An International Multicenter Study. Ann Surg. 2023 Jul 1;278(1):118-126. doi: 10.1097/SLA.0000000000005666. Epub 2022 Aug 11. PMID 35950757
- [Background] Siegel RL, Kratzer TB, Giaquinto AN, Sung H, Jemal A. Cancer statistics, 2025. CA Cancer J Clin. 2025 Jan-Feb;75(1):10-45. doi: 10.3322/caac.21871. Epub 2025 Jan 16. PMID 39817679
- [Background] McGuigan A, Kelly P, Turkington RC, Jones C, Coleman HG, McCain RS. Pancreatic cancer: A review of clinical diagnosis, epidemiology, treatment and outcomes. World J Gastroenterol. 2018 Nov 21;24(43):4846-4861. doi: 10.3748/wjg.v24.i43.4846. PMID 30487695
- [Background] Kleeff J, Korc M, Apte M, La Vecchia C, Johnson CD, Biankin AV, Neale RE, Tempero M, Tuveson DA, Hruban RH, Neoptolemos JP. Pancreatic cancer. Nat Rev Dis Primers. 2016 Apr 21;2:16022. doi: 10.1038/nrdp.2016.22. PMID 27158978